CLINICAL TRIAL: NCT07334678
Title: Early Results of Transanal Opening of the Intersphincteric Space (TROPIS) Versus Coring Out Fistulectomy in Management of High Anal Fistulas: A Randomized Clinical Trial
Brief Title: TROPIS Versus Coring Out Fistulectomy in High Anal Fistula
Acronym: TROCO-HAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelaal, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-311-2025
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: High Anal Fistula
Keywords: TROPIS; Intersphincteric Space; Coring Out Fistulectomy; High anal fistulas; Sphincter-Preserving Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transanal Opening of the Intersphincteric Space (TROPIS) (Experimental): patient with high anal fistula will be treated with Transanal Opening of the Intersphincteric Space (TROPIS)
  Interventions: Procedure: Transanal opening of intersphincteric space (TROPIS)
- Coring Out Fistulectomy (Active Comparator): patient with high anal fistula will be treated with Coring Out Fistulectomy
  Interventions: Procedure: Coring Out Fistulectomy

INTERVENTIONS:
Procedure: Transanal opening of intersphincteric space (TROPIS) — The fistula tracts on both sides of the External anal sphincter (EAS) are separately dealt with. A curved artery forceps is inserted in the fistula tract in the intersphincteric space through the internal opening.The mucosa and the internal sphincter overlying the artery forceps are then incised with electrocautery. The edges of the resulting wound are trimmed and A gutter is made inferiorly from the opened-up intersphincteric space to the anal verge to facilitate drainage from the intersphincteric space wound in the postoperative period.The fistula tract lateral to (outside) the EAS will be excised till the external anal sphincter.
  Arms: Transanal Opening of the Intersphincteric Space (TROPIS)
Procedure: Coring Out Fistulectomy — Incision was made around external opening.Coring out the fistulous track using a combination of cutting and coagulation diathermy from external opening to internal opening with closure of internal opening
  Arms: Coring Out Fistulectomy

SUMMARY:
High anal fistulas represent a surgical challenge due to high recurrence rates and risk of postoperative fecal incontinence. Several sphincter-preserving techniques have been developed to address these issues. Coring Out fistulectomy is a traditional sphincter-saving approach, while Transanal Opening of the Intersphincteric Space (TROPIS) is a recently introduced technique with promising outcomes. This randomized clinical trial aims to compare the efficacy, safety, and patient outcomes of TROPIS versus coring out fistulectomy in the management of high complex anal fistulas.

DETAILED DESCRIPTION:
Fistula-in-ano is an abnormal epithelialized tract connecting the anal canal to the perianal skin, most commonly caused by cryptoglandular infection. High anal fistulas, involving more than one-third of the sphincter complex, carry a significant risk of postoperative incontinence when treated with fistulotomy. As a result, sphincter-preserving techniques have introduced.

Coring out fistulectomy allows excision of the fistulous tract while preserving sphincter integrity but has variable recurrence rates. TROPIS involves transanal opening of the intersphincteric space with complete preservation of the external anal sphincter and has shown high success rates in recent studies.

This prospective randomized clinical trial compares TROPIS and coring out fistulectomy regarding Failure rate (defined as failure of healing or recurrence of anal fistula), operative time, time for wound healing and postoperative complications including fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high anal fistula ( involving more than 1/3 of the sphincter complex), whether de novo or recurrent

Exclusion Criteria:

* Patients with fistula secondary to malignancy, inflammatory bowel disease, trauma or radiation
* Patients with Low anal fistula
* Patient with preoperative fecal incontinence
* Previous levator ani muscle injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Compares Failure rate of TROPIS versus Coring Out fistulectomy in high fistula | Up to 4 months postoperatively
  Compares Failure rate of TROPIS versus Coring Out fistulectomy in high fistula (failure of healing or recurrence of anal fistula), Early results

SECONDARY OUTCOMES:
Operative time | During surgery
  compare time of operation between both procedure
Hospitalization period | From surgery until discharge
  compare how many days patients stay in hospital postoperatively in both groups
surgical site infection | Up to 4 months postoperatively
  compare surgical site infection in both groups
Time for wound Healing | Up to 4 months postoperatively
  Time for wound Healing in both groups
Postoperative bleeding | Up to 4 months postoperatively
  compare Postoperative bleeding in both groups
postoperative fecal incontinence | Up to 4 months postoperatively
  compare post postoperative fecal incontinence in both groups
Time to return to normal activity | Up to 4 months postoperatively
  Compare Time to return to normal activity in both groups
Postoperative urine retention | Within 48 hours postoperatively
  compare postoperative urine retention in both groups
Pain intensity | At day 1 and day 7 postoperatively
  Compare Pain intensity measured using Visual Analogue Scale between both groups (Visual Analogue Scale for Pain: ranges from 0 to 10 . Higher scores indicate a worse outcome {greater pain intensity}).

CONTACTS AND LOCATIONS:
Overall Officials: Haitham M.Azmy Basiouny, Lecturer, Study Director — Cairo University
Locations (1):
- Faculty of medicine Cairo University, Cairo, Al-Manial Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a small surgical trial with a limited number of participants, and sharing raw data could lead to identification of participants